CLINICAL TRIAL: NCT04646187
Title: De-escalation of Anti-TNF Therapy in Adolescents and Young Adults With IBD With Tight Faecal Calprotectin and Trough Level Monitoring
Brief Title: De-escalation of Anti-TNF Therapy in Inflammatory Bowel Disease
Acronym: FREE
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: European Crohn´s and Colitis Organisation (Unknown); Bühlmann Laboratories AG (Industry)
Responsible Party: Principal Investigator, P.F. van Rheenen, MD PhD, University Medical Center Groningen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202000261; 2020-001811-26 (EudraCT Number)
Record Dates: First submitted 2020-11-20; First posted 2020-11-27 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2025-01

CONDITIONS: Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative
Keywords: Infliximab; Adalimumab; Tumor Necrosis Factor-alpha; Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative | interventions — Infliximab; CT-P13; Adalimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): In patients treated with adalimumab, the dosing interval will be lengthened from 2 to 3 weeks. In patients treated with infliximab, the dosing interval will be lengthened from 8 to 12 weeks. Consists of two groups: Patients randomised to the intervention group and patients allocated to the intervention group based on preference.
  Interventions: Biological: Infliximab; Biological: Adalimumab
- Control group (No Intervention): Unchanged dosing interval. Consists of two groups: Patients randomised to the control group and patients allocated to the control group based on preference.

INTERVENTIONS:
Biological: Infliximab — Dosing interval lengthening from 8 to 12 weeks
  Other Names: Remicade; Flixabi; Inflectra; Remsima; Zessly
  Arms: Intervention group
Biological: Adalimumab — Dosing interval lengthening from 2 to 3 weeks
  Other Names: Humira; AMGEVITA; Hulio; Hyrimoz; Idacio; Imraldi
  Arms: Intervention group

SUMMARY:
BACKGROUND/RATIONALE:

Treatment outcomes of patients with inflammatory bowel disease (IBD) have improved enormously during the past decade due to the use of anti-tumour necrosis factor (anti-TNF) therapy. As a result, 67 to 91% of paediatric patients and 66% of adult patients is still in sustained remission two years after the initiation of anti-TNF therapy. Prolonged use of anti-TNFs comes with disadvantages such as dose dependent susceptibility to infections and dermatological adverse effects. Preliminary, mostly uncontrolled studies suggest that dose reduction by dosing interval lengthening is a realistic option in a relevant proportion of patients with IBD, provided that intensive follow-up is applied.

OBJECTIVE:

To evaluate whether a faecal calprotectin (FC) guided strategy of anti-TNF dosing interval lengthening is non-inferior in maintaining remission in patients with IBD, compared with an unchanged dosing interval.

DETAILED DESCRIPTION:
STUDY DESIGN:

International, multi-centre, prospective, partially randomised patient-preference trial.

STUDY POPULATION:

Study population: Eligible patients are aged 12-25 years with luminal Crohn's disease (CD) or ulcerative colitis (UC), who have three consecutive faecal calprotectin (FC) results in the target range (i.e. <250 µg/g for CD patients; <150 µg/g for UC patients) over a period of 6 months at study entry or recently confirmed endoscopic remission.

DE-ESCALATION STRATEGY:

In patients treated with adalimumab, the dosing interval will be lengthened from 2 to 3 weeks. In patients treated with infliximab, the dosing interval will be lengthened from 8 to 12 weeks. FC rapid tests will be performed every 4 weeks and rapid tests for anti-TNF trough levels will be performed every 12 weeks.

MAIN STUDY ENDPOINTS:

The primary outcome is the cumulative incidence of out-of-range FC results at 48 weeks follow-up. Secondary endpoints include time to get out-of-range FC results, cumulative incidence of anti-TNF associated adverse effects, proportion of patients progressing from out-of-range FC to loss-of-response and identification of predictors of successful de-escalation.

ETHICAL CONSIDERATIONS:

Patients with reduced anti-TNF exposure may have a higher risk of out-of-range FC results and, on the other hand, may benefit from fewer hospital visits or injections and possibly a decrease in adverse effects of anti-TNF therapy. Tight monitoring of FC levels (i.e. 4-weekly) will allow institution of re-escalation before the patient manifests clinical signs of relapse. This study cannot be conducted without the participation of minors and young adults, who typically have a short disease duration. Early treatment with anti-TNF agents possibly modifies the course of their disease, which makes provision for safe deescalation.

ELIGIBILITY:
Inclusion Criteria:

* Aged 12-25 years
* Diagnosed with luminal Crohn's disease or ulcerative colitis
* Treated with either 8-weekly infliximab or 2-weekly adalimumab
* Current anti-TNF agent as first ever anti-TNF agent or prior anti-TNF agent discontinued for reason other than primary non-response or secondary loss-of-response
* No previous attempts to lengthen the dosing interval
* Three consecutive faecal calprotectin (FC) results in the target range (i.e. <250 μg/g for CD patients; <150 μg/g for UC patients) in the previous 6 months or confirmed endoscopic remission within 2 months before study entry (i.e. simple endoscopic score for Crohn's disease (SES-CD) <3 points for CD patients; ulcerative colitis endoscopic index of severity (UCEIS) ≤1 point for UC patients)
* Absence of symptoms associated with active IBD (judged by the local IBD-team)
* Written informed consent granted

Exclusion Criteria:

* Perianal fistula
* Presence of ileostomy or ileoanal pouch (as FC cut-off is not validated for small bowel faeces)
* Any inflammatory comorbidity, such as rheumatoid arthritis
* Current treatment with corticosteroids (prednisone or budesonide)
* Current pregnancy

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 148 (Estimated)
Dates: Start 2021-03-11 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
cumulative incidence of out-of-range fecal calprotectin results at 48 weeks follow-up | 48 weeks
  Out-of-range FC results are defined as fecal calprotectin above the target range (i.e. >250 μg/g for CD patients; >150 μg/g for UC patients) and at least 100 μg/g increase compared with the previous result, unless the previous result was already above the target range.

SECONDARY OUTCOMES:
Time to get out-of-range fecal calprotectin results | up to 48 weeks
  The time from study baseline until the first out-of-range fecal calprotectin result
Cumulative incidence of anti-TNF-associated respiratory infections and dermatological adverse effects at 48 weeks follow-up | 48 weeks
  Dermatological adverse effect include skin infections, new-onset or worsening of psoriasis, psoriasiform lesions, eczema, acne and alopecia
Evolution of FC and anti-TNF trough levels in the first 16 weeks after reverting to previous dosing interval | Up to 48+16 weeks
  Proportion of patients with return of FC levels to target range without switch to out-of-class biological
Proportion of patients developing loss-of-response in the first 16 weeks after reverting to the previous dosing interval | Up to 48+16 weeks
  Loss-of-response is defined as the appearance of symptoms of active IBD in combination with persistent out-of-range fecal calprotectin results
Identification of predictors of successful de-escalation. | 48 weeks
  Predictors of successful de-escalation will be assessed by calculating odds ratios with the use of univariate logistic regression analysis. Candidate predictors with p<0.10 in univariate analysis will be selected for use in the multivariate analysis.

OTHER OUTCOMES:
Patients' attitudes towards deprescribing anti-TNF agents | 48 weeks
  We will use the revised Patients' Attitudes Towards Deprescribing (rPATD) questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Patrick F van Rheenen, MD PhD, Principal Investigator — University Medical Center Groningen
Locations (7):
- Belgium (3):
  - Universitair Ziekenhuis Gent, Ghent
  - Centre hospitalier universitaire de Liège, Liège
  - Centre hospitalier régional de la Citadelle, Liège
- Netherlands (3):
  - Rijnstate Hospital, Arnhem
  - Catharina Hospital Eindhoven, Eindhoven
  - University Medical Center Groningen, Groningen
- Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bouhuys M, Lexmond WS, Dijkstra G, Lobaton T, Louis E, van Biervliet S, Groen H, Guardiola J, Rheenen PV. Efficacy of anti-TNF dosing interval lengthening in adolescents and young adults with inflammatory bowel disease in sustained remission (FREE-study): protocol for a partially randomised patient preference trial. BMJ Open. 2021 Nov 3;11(11):e054154. doi: 10.1136/bmjopen-2021-054154. PMID 34732500